CLINICAL TRIAL: NCT03153956
Title: A Prospective, Randomized Double-Armed Efficacy Evaluation of AposTherapy® for the Treatment of Knee Osteoarthritis
Brief Title: Efficacy of AposTherapy® in Knee OA
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Halt in funding
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14-02127
Record Dates: First submitted 2017-05-09; First posted 2017-05-15 (Actual); Results first posted 2020-03-24 (Actual); Last update posted 2020-03-24 (Actual); Status verified 2020-03

CONDITIONS: Osteoarthritis, Knee
Keywords: AposTherapy® System; Osteoarthritis; Total knee arthroplasties; Degenerative joint disease
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis; Joint Diseases

STUDY DESIGN:
Intervention Model Description: Phase I - A prospective, interventional, randomized, double-arm clinical evaluation of patients who have been diagnosed with OA of the knee. The active treatment arm (personally calibrated biomechanical device) will be compared to a control arm (sham-placebo device) (similar shoes without biomechanical elements).
  Phase II - Open-label, cross-over study design. After the completion of phase one patients will be un-blinded to their group allocation. Patients that were allocated to the sham-placebo control group will cross to the active group and will receive the AposTherapy treatment. Patients that were allocated to the active group will continue with treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Active Treatment Arm (Experimental): Personally calibrated bio-mechanical device
  Interventions: Device: Calibrated AposTherapy®
- Control Arm (Placebo Comparator): sham-placebo device (similar shoes without bio-mechanical elements).
  Interventions: Device: Non-Calibrated Sham Apos Therapy Device

INTERVENTIONS:
Device: Calibrated AposTherapy® — a biomechanical device including 2 hemispheric biomechanical elements attached to a platform in a form of a shoe. the biomechanical device is calibrated to each patient by a physiotherapist specialized with the treatment methodology.
  Arms: Active Treatment Arm
Device: Non-Calibrated Sham Apos Therapy Device — The comparator group will receive a non-calibrated sham device.
  Arms: Control Arm

SUMMARY:
A prospective, interventional, randomized, double-arm clinical evaluation study to examine the efficacy of AposTherapy® versus a control group, in the short-term at 6 months and in the long-term at 12 months post-treatment, with the primary efficacy assessment based on improvement in knee pain score and improvement in function in patients following diagnosis of knee osteoarthritis (OA).

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from symptomatic unilateral or bilateral knee OA at the medial compartment for at least six months;
* Fulfilling the ACR clinical criteria;
* Having radiographically assessed OA of the knee with a Kellgren-Lawrence grade more than or equal to grade 2; and,
* Having VAS-Pain ≥ 3, on a scale between 0-10.
* Patients who have a shoe size between US 4 and US 12

Exclusion Criteria:

* Patients suffering from acute septic arthritis.
* Patients who received a corticosteroid injection within 3 months of the study.
* Patients who received hyaluronic acid (HA) injections within 6 months of the study
* Patients suffering from avascular necrosis of the knee.
* Patients with a history of knee buckling or recent knee injury.
* Patients who have had a joint replacement or other major surgery to the knee, hip or ankle (ipsilateral or contralateral side).
* Patients suffering from neuropathic arthropathy.
* Patients with an increased tendency to fall.
* Patients exhibiting a lack of physical or mental ability to perform or comply with the study procedure.
* Patients with a history of pathological osteoporotic fracture.
* Patients suffering from symptomatic degenerative arthritis in lower limb joints other than the knees.
* Patients with referred pain in the knees from primary back or hip joint pain.
* Patients with neurological deficits to the lower extremity (ex. foot drop)
* Patients whose shoe size is less than US 4 and greater than US 12
* Patients who have had arthroscopy within 6 months of the study
* Patients with inflammatory arthropathy

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2015-04-16 (Actual); Primary Completion 2018-11-15 (Actual); Study Completion 2018-11-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Cardone, DO, Principal Investigator — NYU Langone Health
Locations (1):
- New York University School of Medicine, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Active Treatment Arm | Control Arm
Started | 39 | 38
Completed | 39 | 38
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Treatment Arm | Control Arm | Total
Number analyzed (Participants) | 39 | 38 | 77
Age, Continuous [Mean (Standard Deviation); unit: years] | 62 (9) | 61 (8.2) | 61 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 27 | 54
  Male | 12 | 11 | 23
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Western Ontario and McMaster University (WOMAC) Total Score
Description: WOMAC evaluates the condition of patients with osteoarthritis of the knee and hip, including pain, stiffness, and physical functioning of the joints. In this study, WOMAC scores were recomputed as the sum within sub-scales (pain score is the sum of questions 1-5; stiffness is the sum of questions 6-7; functional score is the sum of questions 8-24). The total score is reported as the sum of the pain, stiffness, and functional sub-scores for all participants. The total score range is 0-1292. Higher scores on the WOMAC indicate worse pain, stiffness, and functional limitations.
Time Frame: screening, 3 months, 6 months, 9 months, and 12 months
Population: Participants who scheduled visits beyond 4 days before or after the specified timeframes (3, 6, and 9 months from screening) were not included in the analysis. (Treatment participants did not have a 9 month visit)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Treatment Arm | Control Arm
Number analyzed (Participants) | 38 | 34
score on a scale
  WOMAC Total score - screen | 1062.7 (545.96) | 975.1 (580.87)
  WOMAC Total score - 3 months: number analyzed (Participants) | 27 | 23
  WOMAC Total score - 3 months | 548.8 (440.22) | 601.1 (467.39)
  WOMAC Total Score - 6 months: number analyzed (Participants) | 21 | 22
  WOMAC Total Score - 6 months | 420.2 (391.7) | 524.8 (448.83)
  WOMAC Total Score - 9 months: number analyzed (Participants) | 0 | 11
  WOMAC Total Score - 9 months |  | 280.2 (194.84)
  WOMAC Total Score - 12 months: number analyzed (Participants) | 14 | 10
  WOMAC Total Score - 12 months | 396.5 (324.99) | 433 (352.32)

2. Secondary Outcome: Visual Analog Score (VAS) Score
Description: The visual analogue scale or visual analog scale (VAS) is a psychometric response scale which can be used in questionnaires. It is a measurement instrument for subjective characteristics or attitudes that cannot be directly measured.
Time Frame: 12 Months
Population: Data was not collected for this outcome measure due to study termination.
Arm/Group | Active Treatment Arm | Control Arm
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Short-Form 36 (SF-36) Total Score
Description: The Short Form (36) Health Survey is a 36-item, patient-reported survey of patient health. The survey consists eight scaled scores; the scores are weighted sums of the questions in each section. Scores range from 0-100, with lower scores = more disability and higher scores = less disability. Therefore, higher scores represent better health.
Time Frame: screening, 3 months, 6 months, 9 months, and 12 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Treatment Arm | Control Arm
Number analyzed (Participants) | 38 | 37
score on a scale
  SF-36 total score - screening | 55.6 (15.03) | 56.6 (16.77)
  SF-36 total score - 3 months: number analyzed (Participants) | 27 | 23
  SF-36 total score - 3 months | 64.6 (16.8) | 63.0 (17.09)
  SF-36 total score - 6 months: number analyzed (Participants) | 21 | 21
  SF-36 total score - 6 months | 69.7 (14.8) | 68 (17.21)
  SF-36 total score - 9 months: number analyzed (Participants) | 0 | 11
  SF-36 total score - 9 months |  | 74.5 (6.37)
  SF-36 total score - 12 month: number analyzed (Participants) | 14 | 10
  SF-36 total score - 12 month | 71 (9.77) | 66.6 (15.38)

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Active Treatment Arm | Control Arm
All-Cause Mortality (participants affected / at risk) | 0/39 | 0/38
Serious Adverse Events (participants affected / at risk) | 0/39 | 0/38
Other Adverse Events (participants affected / at risk) | 0/39 | 0/38

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-06-23): https://cdn.clinicaltrials.gov/large-docs/56/NCT03153956/Prot_SAP_000.pdf